CLINICAL TRIAL: NCT04412616
Title: A Phase 1, Multicenter, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Preliminary Evidence of Antitumor Activity of ZZ06 in Adult Patients With Advanced Solid Tumor Malignancies
Brief Title: ZZ06 in Adult Patients With Advanced Solid Tumor Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun Intellicrown Pharmaceutical Co. LTD (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZZ06-2020A
Record Dates: First submitted 2020-05-14; First posted 2020-06-02 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Advanced EGFR Positive Solid Tumor
Keywords: treatment-emergent adverse event (TEAE); dose limiting toxicity (DLT); pharmacokinetic (PK); antidrug antibodies (ADA)

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- ZZ06 0.03 mg/kg dose group (Experimental): ZZ06 0.03 mg/kg will be administered twice weekly.A cycle is defined as continuous treatment for 28 days, and the initial treatment course is 2 cycles. Patients can receive up to 6 additional cycles unless disease progression, unacceptable toxicity, or other protocol specified stopping criteria occur. After 6 cycles, additional cycles may be given upon request by the Investigator and approval by the Medical Monitor.
  Interventions: Biological: ZZ06
- ZZ06 0.06 mg/kg dose group (Experimental): ZZ06 0.06 mg/kg will be administered twice weekly.A cycle is defined as continuous treatment for 28 days, and the initial treatment course is 2 cycles. Patients can receive up to 6 additional cycles unless disease progression, unacceptable toxicity, or other protocol specified stopping criteria occur. After 6 cycles, additional cycles may be given upon request by the Investigator and approval by the Medical Monitor.
  Interventions: Biological: ZZ06
- ZZ06 0.12 mg/kg dose group (Experimental): ZZ06 0.12 mg/kg will be administered twice weekly.A cycle is defined as continuous treatment for 28 days, and the initial treatment course is 2 cycles. Patients can receive up to 6 additional cycles unless disease progression, unacceptable toxicity, or other protocol specified stopping criteria occur. After 6 cycles, additional cycles may be given upon request by the Investigator and approval by the Medical Monitor.
  Interventions: Biological: ZZ06
- ZZ06 0.22 mg/kg dose group (Experimental): ZZ06 0.22 mg/kg will be administered twice weekly.A cycle is defined as continuous treatment for 28 days, and the initial treatment course is 2 cycles. Patients can receive up to 6 additional cycles unless disease progression, unacceptable toxicity, or other protocol specified stopping criteria occur. After 6 cycles, additional cycles may be given upon request by the Investigator and approval by the Medical Monitor.
  Interventions: Biological: ZZ06
- ZZ06 0.39 mg/kg dose group (Experimental): ZZ06 0.39 mg/kg will be administered twice weekly.A cycle is defined as continuous treatment for 28 days, and the initial treatment course is 2 cycles. Patients can receive up to 6 additional cycles unless disease progression, unacceptable toxicity, or other protocol specified stopping criteria occur. After 6 cycles, additional cycles may be given upon request by the Investigator and approval by the Medical Monitor.
  Interventions: Biological: ZZ06
- ZZ06 0.70 mg/kg dose group (Experimental): ZZ06 0.70 mg/kg will be administered twice weekly.A cycle is defined as continuous treatment for 28 days, and the initial treatment course is 2 cycles. Patients can receive up to 6 additional cycles unless disease progression, unacceptable toxicity, or other protocol specified stopping criteria occur. After 6 cycles, additional cycles may be given upon request by the Investigator and approval by the Medical Monitor.
  Interventions: Biological: ZZ06
- ZZ06 1.00 mg/kg dose group (Experimental): ZZ06 1.00 mg/kg will be administered twice weekly.A cycle is defined as continuous treatment for 28 days, and the initial treatment course is 2 cycles. Patients can receive up to 6 additional cycles unless disease progression, unacceptable toxicity, or other protocol specified stopping criteria occur. After 6 cycles, additional cycles may be given upon request by the Investigator and approval by the Medical Monitor.
  Interventions: Biological: ZZ06

INTERVENTIONS:
Biological: ZZ06 — The phase I "3 + 3" study design was used in dose escalation from low dose to high dose to determine the MTD.Sequential assignment of Patient cohorts to one of five dose levels of ZZ06 : 0.03mg/kg,0.06mg/kg,0.12mg/kg,0.22mg/kg,0.39mg/kg,0.70mg/kg,1 mg/kg.

SUMMARY:
This is a Phase 1, Multicenter, Open-label study to assess the safety, tolerability and preliminary efficacy of ZZ06 in participants with all Adult Patients with Advanced EGFR-positive Solid Tumor Malignancies who are not able to have current standard anti-tumor therapies. The purpose of this study is to determine the maximum tolerated dose (MTD) , to characterise the safety, pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD) and anti-tumor activity of ZZ06 as a single agent in adult participants with advanced solid tumors.

DETAILED DESCRIPTION:
The study will start with an accelerated-titration dose escalation scheme, enrolling 1 patient per cohort for the first 2 cohorts with expansion to 3 patients in the event of Grade ≥ 2 treatment-emergent adverse event (TEAE) or dose limiting toxicity (DLT) possibly, probably, or definitely related to the study drug. After the first 2 cohorts, the study will then proceed to a 3+3 design, with enrollment of 3 patients per cohort and expansion to 6 patients in the event of a DLT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed advanced solid tumor that is positive for EGFR and has progressed despite standard therapy or for whom no standard therapy exists.
* Patients are required to have archival tumor tissue available for assessment of EGFR status via FDA-approved EGFR assay .
* Age ≥ 18 years.
* Patients must have at least 1 measurable lesion as defined by RECIST v1.1.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Life expectancy ≥ 12 weeks.
* Baseline organ function and laboratory data meet the following criteria:

  1. Bone marrow： ANC ≥ 1500 cells/mm3； Platelet count ≥ 75 000 cells/mm3； Hemoglobin ≥ 8.0 g/dL.
  2. Coagulation： Prothrombin time ≤ 1.5× ULN； Activated partial thromboplastin time ≤ 1.5× ULN；
  3. Renal function： Serum creatinine ≤ 1.5× ULN ； estimated glomerular filtration rate≥ 60 mL/min (Cockcroft-Gault formula).
  4. Hepatic function： Serum total bilirubin ≤ 1.5 mg/dL； AST and ALT ≤ 3.0× ULN (if metastases are present, ≤ 5.0× ULN).
* Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.Patients must provide written informed consent prior to any study procedures.

Exclusion Criteria:

* History of another primary cancer ≤ 3 years, with the exception of completely resected nonmelanoma skin cancer or carcinoma in situ of uterine cervix.
* Active or symptomatic CNS metastases. Patients with treated CNS metastases that have been stable for ≥ 4 weeks and do not require treatment with steroids or anticonvulsants may be enrolled at the discretion of the Investigator.
* Tests positive for hepatitis C virus, hepatitis B virus, or human immunodeficiency virus infection.
* Active, clinically significant infections.
* Clinically significant cardiovascular disease, including any of the following:

  1. Congestive heart failure (New York Heart Association Class > 2).
  2. Serious cardiac arrhythmia.
  3. Myocardial infarction ≤ 6 months.
  4. Unstable angina.
* Prior clinically significant allergic reaction to chimerized or murine monoclonal antibody therapy.
* Prior treatment ≤ 6 months with cetuximab, panitumomab, gefitinb, erlotinib, or other therapy that specifically and directly targets the EGF pathway.
* Anticancer therapy or investigational agents for nonmalignant disease ≤ 4 weeks or 5 half-lives, whichever is shorter, prior to Cycle 1 Day 1, with the exception of tamoxifen for patients with a history of operated breast cancer > 3 years and no evidence of disease after surgery.
* Major surgery ≤ 4 weeks.
* Clinically significant psychiatric illness, other comorbidity, or laboratory abnormality that, in the opinion of the Investigator, makes it unsafe for the patient to participate in the study or may interfere with study compliance or study results.
* Other unspecified reasons that, in the opinion of the Investigator, make the patient unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-06 (Estimated)

PRIMARY OUTCOMES:
ZZ06 AEs | up to 36 weeks
  Adverse events will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events v5.0
Incidence of abnormal laboratory test results | up to 36 weeks
  The data of the clinical laboratory evaluation is collected and analyzed according to the time point of the test flow chart
Incidence of abnormal physical exam findings | up to 36 weeks
  The data of the physical examinations is collected and analyzed according to the time point of the test flow chart

SECONDARY OUTCOMES:
PK parameters: Area under curve (AUC) | up to 28 weeks
  According to the test schedule, the blood volume of each subject's PK was analyzed and PK analysis was performed.
PK parameters: Cmax | up to 28 weeks
  According to the test schedule, the blood volume of each subject's PK was analyzed and PK analysis was performed.
PK parameters: Clearance rate (CL) | up to 28 weeks
  According to the test schedule, the blood volume of each subject's PK was analyzed and PK analysis was performed.
PK parameters: t1/2 | up to 28 weeks
  According to the test schedule, the blood volume of each subject's PK was analyzed and PK analysis was performed.
PK parameters: Vz | up to 28 weeks
  According to the test schedule, the blood volume of each subject's PK was analyzed and PK analysis was performed.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Goel, MD, Principal Investigator — Montefiore Medical Center
Locations (5):
- United States (3):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kansas University Cancer Center, Fairway, Kansas
  - Montefiore Medical Center, The Bronx, New York
- China (2):
  - Jilin Cancer Hospital, Changchun, Jilin
  - The first Bethune hospital of Jilin University, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: No